CLINICAL TRIAL: NCT05524246
Title: Pilot Trial of Pravastatin as a Novel Prophylactic Medicine to Reduce Endothelial Injury in Pediatric Patients With Elevated Body Mass Index
Brief Title: Pravastatin as a Prophylactic to Reduce Endothelial Injury in Pediatric Patients With Elevated Body Mass Index
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0308
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Stem Cell Transplant (HSCT); Endothelial Injury
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pravastatin Prophylactic Treatment (Experimental)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Participants will receive pravastatin orally once daily through the first 35 days after bone marrow transplant.

SUMMARY:
Chemotherapy and radiation used in patients undergoing bone marrow transplant (BMT) disrupts the endothelial lining (a thin layer of cells inside the blood vessels) which is found all throughout the body including the kidney, heart, lungs, and intestines. Disruption of this endothelial lining can lead to complications such as graft-vs-host disease (GVHD), thrombotic microangiopathy (TMA) and veno-occlusive disease (VOD). The purpose of this research study is to help investigators see if pravastatin is safe and well tolerated in patients undergoing BMT to see if it will reduce endothelial injury after BMT.

The investigator hypothesizes that prophylactic pravastatin in pediatric allogeneic hematopoietic stem cell transplant recipients with elevated BMI is safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for allogeneic stem cell transplant
* Ages ≥ 2 - ≤ 25 years old
* Elevated BMI defined by the Center for Disease Control and Prevention definitions. Both overweight (BMI between 85th-94th percentile) and obese (BMI >95th percentile) patients are eligible
* All diagnoses are eligible

Exclusion Criteria:

* Patients with documented anaphylaxis to pravastatin
* Patients will be ineligible if they are unable to take medication orally or enterally (i.e. intestinal failure)
* Patients with elevations in ALT/AST levels 3x ULN at time of enrollment
* Patients with renal impairment as clinically measured (GFR <50 ml/min/1.73m2) at time of enrollment
* Patients with known neuromuscular and metabolic disorders associated with an increased risk of rhabdomyolysis (ie metabolic muscle disorders, mitochondrial disorders, and muscular dystrophies)
* Patients taking any drugs that are known substrates for OATP1B1 and OATP1B3 transporters

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who developed clinically significant transaminitis, renal dysfunction and rhabdomyolysis | Until day 35 after bone marrow transplant when pravastatin is discontinued
  Every enrolled patient will have routine liver function test (LFT) and renal function profile monitoring as part of their standardized transplant care. Transaminitis is expected and often multifactorial in the HSCT population, (i.e. preparative regimen, azole antifungal prophylaxis, or post-transplant complications such as infection and GVHD), therefore, we have determined modified parameters to hold or modify the dose of pravastatin. We will modify and/or hold pravastatin dosing at the time of transaminase elevations > 3X upper limit of normal unless a clear-cut alternative explanation can be provided. Additionally, we will also check creatinine kinase (CK) levels on admission and once weekly while the patient is actively taking pravastatin to monitor for rhabdomyolysis.
Percentage of participants who adhered to the medication plan | Until day 35 after bone marrow transplant when pravastatin is discontinued
  Participants will be considered adhered to the medication plan if they took the study drug at least 70% of the time. Nursing documentation of pravastatin administration and drug diaries will be used as documentation of compliance.

SECONDARY OUTCOMES:
Number of participants with overall survival | 100 days after bone marrow transplant
Number of participants with graft failure | 100 days after bone marrow transplant
  Graft failure is defined as follows:
  Primary graft failure is defined as no evidence of engraftment or hematological recovery of donor cells, within the first month after transplant, without evidence of disease relapse.
  Secondary graft failure refers to the loss of a previously functioning graft, resulting in cytopenia involving at least two blood cell lineages.
Number of participants with primary disease relapse | 100 days after bone marrow transplant
  Primary disease relapse is defined as: The return of a disease or the signs and symptoms of a disease after a period of improvement.
Median number of days until neutrophil engraftment | Through study completion, an average of up to 100 days
  Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm3 (0.5 x 10^9/L) or greater.
Median number of days until platelet engraftment | Through study completion, an average of up to 100 days
  Platelet engraftment is usually defined as independence from platelet transfusion for at least 7 days with a platelet count of more than >20 × 10^9/L
Assessment of SLCO1B1 genotyping | Baseline
  The SLCO1B1 gene encodes for making the protein organic anion transporting polypeptide 1B1 (OATP1B1), which is the transporter for drugs, including statins, into the liver. Patients enrolled on study will have their SLCO1B1 genotyping performed from whole blood samples at baseline to determine how this affects their overall statin clearance.
Measurement of sphingosine-1-phosphate (S1P) levels in plasma | Weekly from admission until day 35 from bone marrow transplant
  S1P levels will be measured on weekly intervals using mass spectrometry
Number of participants who adhered to the medication plan | Through study completion, an average of 35 days after bone marrow transplant
  The lipid profile is a blood test that includes measurements of cholesterol, triglycerides, High-density lipoprotein (HDL) and Low-density lipoprotein (LDL). It is a routine test that monitors cholesterol levels. Pravastatin reduces cholesterol production. The lipid profile will be measured prior to the first dose of pravastatin. After the last dose of pravastatin the lipid profile will be measured. Any reduction in total cholesterol and LDL levels will be used as a surrogate marker for medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Koo, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States